CLINICAL TRIAL: NCT01342796
Title: A Phase II, Randomized, Controlled, Observer-Blind, Clinical Study to Evaluate the Humoral and Cell Mediated Immunity and Safety of Two Intramuscular Doses of MF59C.1-adjuvanted Subunit Influenza Vaccine or Conventional Subunit Influenza Vaccine in Previously Unvaccinated Healthy Subjects Aged 6 to <36 Months
Brief Title: Humoral and Cell Mediated Immunity and Safety of MF59C.1-adjuvanted Subunit Influenza Vaccine or a Conventional Subunit Influenza Vaccine in Previously Unvaccinated Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V70_34; 2010-023791-63 (EudraCT Number)
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2019-02

CONDITIONS: Seasonal Influenza; Influenza; Influenza Due to Unspecified Influenza Virus; Human Influenza
Keywords: Cell mediated immunity; cell mediated immune response; Children; adjuvanted
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Biological: MF59C.1-adjuvanted subunit influenza vaccine
- Arm 2 (Active Comparator)
  Interventions: Biological: Sub unit, Inactivated, Influenza vaccine

INTERVENTIONS:
Biological: MF59C.1-adjuvanted subunit influenza vaccine — 2 x 0.25 ml doses administered intramuscularly in the deltoid muscle of (preferably) the non dominant arm
  Arms: Arm 1
Biological: Sub unit, Inactivated, Influenza vaccine — 2 x 0.25 ml doses administered intramuscularly in the deltoid muscle of (preferably) the non dominant arm
  Arms: Arm 2

SUMMARY:
This study aims to evaluate the immunogenicity, by means of cell mediated immunity (CMI) and hemagglutination inhibition (HI) assay, and also the safety of a MF59C.1-adjuvanted subunit influenza vaccine compared with a conventional subunit vaccine in previously unvaccinated children aged 6 to <36 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and female previously unvaccinated healthy children aged 6 to <36 months.

Exclusion Criteria:

* Any known or suspected impairment of the immune system, any serious disease.
* Any subjects receiving licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
* Individuals who have had influenza vaccine or documented suspected influenza disease prior to day 1.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Site 21: GZA campus Sint Vincentius, Antwerp
  - Site 22: Kinderartsenpraktijk, Hasselt

REFERENCES:
- [Derived] Zedda L, Forleo-Neto E, Vertruyen A, Raes M, Marchant A, Jansen W, Clouting H, Arora A, Beatty ME, Galli G, Del Giudice G, Castellino F. Dissecting the immune response to MF59-adjuvanted and nonadjuvanted seasonal influenza vaccines in children less than three years of age. Pediatr Infect Dis J. 2015 Jan;34(1):73-8. doi: 10.1097/INF.0000000000000465. PMID 25037034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from two sites in Belgium.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- aTIV Group: Subjects received two doses (0.25mL) of MF59C.1-adjuvanted subunit influenza vaccine administered four weeks apart.
- TIV Group: Subjects received two doses (0.25mL) of inactivated, subunit influenza vaccine administered four weeks apart.
Period: Overall Study
Arm/Group | aTIV Group | TIV Group
Started | 43 | 41
Completed | 40 | 38
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 3
Not completed — Inappropriate enrollment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | aTIV Group | TIV Group | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.2 (8.5) | 21.4 (9.7) | 20.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 14 | 34
  Male | 23 | 27 | 50

OUTCOME MEASURES:

1. Primary Outcome: Cell Mediated Immune (CMI) Responses After In-vitro Restimulation Of Peripheral Blood Mononuclear Cells (PBMC) Following Vaccination.
Description: The CMI responses were determined by intracellular staining/Fluorescence-Activated Cell Sorting(ICS/FACS) after in-vitro restimulation of PBMC with vaccine antigens on day 0 and day 50.
Time Frame: Day 1, Day 50
Population: Per Protocol Set
Measure: Mean (95% Confidence Interval); unit: Cells per Million Total Cells
Groups:
- aTIV Group: Subjects received two doses of MF59C.1-adjuvanted subunit influenza vaccine administered four weeks apart.
- TIV Group: Subjects received two doses of inactivated, subunit influenza vaccine administered four weeks apart.
Arm/Group | aTIV Group | TIV Group
Number analyzed (Participants) | 25 | 31
Cells per Million Total Cells
  Any Cytokine - A/H1N1, Day 1: number analyzed (Participants) | 24 | 25
  Any Cytokine - A/H1N1, Day 1 | 631 [477 to 784] | 655 [503 to 806]
  Any Cytokine - A/H1N1, Day 50: number analyzed (Participants) | 24 | 25
  Any Cytokine - A/H1N1, Day 50 | 1560 [1244 to 1876] | 1137 [826 to 1449]
  Any Cytokine - A/H3N2, Day 1 | 503 [346 to 660] | 462 [322 to 602]
  Any Cytokine - A/H3N2, Day 50 | 1328 [1105 to 1550] | 671 [474 to 869]
  Any Cytokine - B/Brisbane, (N=19, 24), Day 1: number analyzed (Participants) | 19 | 24
  Any Cytokine - B/Brisbane, (N=19, 24), Day 1 | 648 [452 to 844] | 753 [579 to 927]
  Any Cytokine - B/Brisbane, Day 50: number analyzed (Participants) | 19 | 24
  Any Cytokine - B/Brisbane, Day 50 | 2369 [1940 to 2798] | 1062 [677 to 1446]
  Any cytokine - B/Florida, Day 1: number analyzed (Participants) | 9 | 18
  Any cytokine - B/Florida, Day 1 | 605 [215 to 996] | 749 [483 to 1015]
  Any cytokine - B/Florida, Day 50: number analyzed (Participants) | 9 | 18
  Any cytokine - B/Florida, Day 50 | 1607 [1113 to 2100] | 996 [662 to 1330]
  Any Cytokine - SEB, Day 1: number analyzed (Participants) | 10 | 17
  Any Cytokine - SEB, Day 1 | 77048 [55913 to 98182] | 107200 [91682 to 122719]
  Any Cytokine - SEB, Day 50: number analyzed (Participants) | 10 | 17
  Any Cytokine - SEB, Day 50 | 80400 [56864 to 103935] | 105013 [88270 to 121755]
  Any cytokine -Tetanus toxoid, Day 1: number analyzed (Participants) | 10 | 16
  Any cytokine -Tetanus toxoid, Day 1 | 1246 [639 to 1852] | 1368 [914 to 1822]
  Any cytokine -Tetanus toxoid, Day 50: number analyzed (Participants) | 10 | 16
  Any cytokine -Tetanus toxoid, Day 50 | 1162 [759 to 1565] | 1229 [928 to 1531]
  IL-2- A/H1N1, Day 1: number analyzed (Participants) | 24 | 25
  IL-2- A/H1N1, Day 1 | 283 [207 to 359] | 240 [165 to 315]
  IL-2- A/H1N1, Day 50: number analyzed (Participants) | 24 | 25
  IL-2- A/H1N1, Day 50 | 1141 [858 to 1423] | 642 [366 to 918]
  IL-2 - A/H3N2, Day 1 | 212 [140 to 283] | 184 [121 to 248]
  IL-2 - A/H3N2, Day 50 | 925 [723 to 1126] | 387 [208 to 566]
  IL-2- B/Brisbane, Day 1: number analyzed (Participants) | 19 | 24
  IL-2- B/Brisbane, Day 1 | 301 [183 to 419] | 330 [225 to 435]
  IL-2- B/Brisbane, Day 50: number analyzed (Participants) | 19 | 24
  IL-2- B/Brisbane, Day 50 | 1704 [1321 to 2087] | 610 [267 to 954]
  IL-2 - B/Florida, Day 1: number analyzed (Participants) | 9 | 18
  IL-2 - B/Florida, Day 1 | 375 [119 to 632] | 275 [100 to 449]
  IL-2 - B/Florida, Day 50: number analyzed (Participants) | 9 | 18
  IL-2 - B/Florida, Day 50 | 1094 [691 to 1497] | 541 [268 to 813]
  IL-2 - SEB, Day 1: number analyzed (Participants) | 10 | 17
  IL-2 - SEB, Day 1 | 67524 [47735 to 87313] | 93312 [78781 to 107843]
  IL-2 - SEB, Day 50: number analyzed (Participants) | 10 | 17
  IL-2 - SEB, Day 50 | 67357 [46682 to 88033] | 92489 [77768 to 107210]
  IL-2 - Tetanus toxoid, Day 1: number analyzed (Participants) | 10 | 16
  IL-2 - Tetanus toxoid, Day 1 | 604 [309 to 899] | 672 [451 to 892]
  IL-2 - Tetanus toxoid, Day 50: number analyzed (Participants) | 10 | 16
  IL-2 - Tetanus toxoid, Day 50 | 659 [291 to 1027] | 765 [489 to 1041]
  IFN-γ - A/H1N1, Day 1: number analyzed (Participants) | 24 | 25
  IFN-γ - A/H1N1, Day 1 | 92 [49 to 135] | 116 [73 to 158]
  IFN-γ - A/H1N1, Day 50: number analyzed (Participants) | 24 | 25
  IFN-γ - A/H1N1, Day 50 | 257 [163 to 350] | 248 [156 to 340]
  IFN-γ - A/H3N2, Day 1 | 78 [44 to 112] | 78 [48 to 108]
  IFN-γ - A/H3N2, Day 50 | 191 [113 to 268] | 130 [61 to 199]
  IFN-γ -B/Brisbane, Day 1: number analyzed (Participants) | 19 | 24
  IFN-γ -B/Brisbane, Day 1 | 83 [37 to 130] | 122 [81 to 163]
  IFN-γ -B/Brisbane, Day 50: number analyzed (Participants) | 19 | 24
  IFN-γ -B/Brisbane, Day 50 | 331 [201 to 462] | 106 [-12.1 to 224]
  IFN-γ - B/Florida, Day 1: number analyzed (Participants) | 9 | 18
  IFN-γ - B/Florida, Day 1 | 112 [46 to 179] | 94 [49 to 139]
  IFN-γ - B/Florida, Day 50: number analyzed (Participants) | 9 | 18
  IFN-γ - B/Florida, Day 50 | 193 [67 to 320] | 145 [59 to 230]
  IFN-γ - SEB, Day 1: number analyzed (Participants) | 10 | 17
  IFN-γ - SEB, Day 1 | 3615 [2110 to 5120] | 4780 [3675 to 5885]
  IFN-γ - SEB, Day 50: number analyzed (Participants) | 10 | 17
  IFN-γ - SEB, Day 50 | 3858 [2367 to 5349] | 4519 [3390 to 5649]
  IFN-γ - Tetanus toxoid, Day 1: number analyzed (Participants) | 10 | 16
  IFN-γ - Tetanus toxoid, Day 1 | 156 [64 to 248] | 148 [80 to 217]
  IFN-γ - Tetanus toxoid, Day 50: number analyzed (Participants) | 10 | 16
  IFN-γ - Tetanus toxoid, Day 50 | 74 [4 to 144] | 163 [10 to 215]
  TNF-α- A/H1N1, Day 1: number analyzed (Participants) | 24 | 25
  TNF-α- A/H1N1, Day 1 | 128 [87 to 170] | 133 [92 to 174]
  TNF-α- A/H1N1, Day 50: number analyzed (Participants) | 24 | 25
  TNF-α- A/H1N1, Day 50 | 495 [368 to 621] | 290 [165 to 415]
  TNF-α - A/H3N2, Day 1 | 81 [56 to 106] | 69 [46 to 91]
  TNF-α - A/H3N2, Day 50 | 447 [324 to 571] | 202 [93 to 311]
  TNF-α - B/Brisbane, Day 1: number analyzed (Participants) | 19 | 24
  TNF-α - B/Brisbane, Day 1 | 116 [62 to 170] | 152 [104 to 200]
  TNF-α - B/Brisbane, Day 50: number analyzed (Participants) | 19 | 24
  TNF-α - B/Brisbane, Day 50 | 921 [658 to 1184] | 251 [13 to 490]
  TNF-α - B/Florida, Day 1: number analyzed (Participants) | 9 | 18
  TNF-α - B/Florida, Day 1 | 149 [50 to 249] | 171 [103 to 238]
  TNF-α - B/Florida, Day 50: number analyzed (Participants) | 9 | 18
  TNF-α - B/Florida, Day 50 | 614 [372 to 857] | 244 [77 to 410]
  TNF-α-SEB, Day 1: number analyzed (Participants) | 10 | 17
  TNF-α-SEB, Day 1 | 25467 [15528 to 35406] | 37856 [30559 to 45154]
  TNF-α-SEB, Day 50: number analyzed (Participants) | 10 | 17
  TNF-α-SEB, Day 50 | 32510 [22453 to 42566] | 34805 [27557 to 42054]
  TNF-α-Tetanus toxoid, Day 1: number analyzed (Participants) | 10 | 16
  TNF-α-Tetanus toxoid, Day 1 | 537 [278 to 795] | 541 [348 to 735]
  TNF-α-Tetanus toxoid, Day 50: number analyzed (Participants) | 10 | 16
  TNF-α-Tetanus toxoid, Day 50 | 384 [156 to 612] | 644 [473 to 815]
  IL-13 - A/H1N1, Day 1: number analyzed (Participants) | 24 | 25
  IL-13 - A/H1N1, Day 1 | 232 [132 to 332] | 170 [71 to 268]
  IL-13 - A/H1N1, Day 50: number analyzed (Participants) | 24 | 25
  IL-13 - A/H1N1, Day 50 | 242 [105 to 378] | 347 [212 to 483]
  IL-13 - A/H3N2, Day 1 | 250 [154 to 346] | 174 [89 to 259]
  IL-13 - A/H3N2, Day 50 | 361 [229 to 494] | 231 [114 to 348]
  IL-13 - B/Brisbane, Day 1: number analyzed (Participants) | 19 | 24
  IL-13 - B/Brisbane, Day 1 | 184 [59 to 308] | 168 [57 to 278]
  IL-13 - B/Brisbane, Day 50: number analyzed (Participants) | 19 | 24
  IL-13 - B/Brisbane, Day 50 | 346 [228 to 463] | 221 [116 to 326]
  IL-13 - B/Florida, Day 1: number analyzed (Participants) | 9 | 18
  IL-13 - B/Florida, Day 1 | 150 [-27.62 to 329] | 88 [-33.78 to 209]
  IL-13 - B/Florida, Day 50: number analyzed (Participants) | 9 | 18
  IL-13 - B/Florida, Day 50 | 97 [18 to 175] | 93 [39 to 146]
  IL-13 -SEB, Day 1: number analyzed (Participants) | 10 | 17
  IL-13 -SEB, Day 1 | 1017 [547 to 1487] | 950 [605 to 1295]
  IL-13 -SEB, Day 50: number analyzed (Participants) | 10 | 17
  IL-13 -SEB, Day 50 | 772 [391 to 1153] | 993 [714 to 1272]
  IL-13 -Tetanus toxoid, Day 1: number analyzed (Participants) | 10 | 16
  IL-13 -Tetanus toxoid, Day 1 | 166 [-0.845 to 333] | 222 [98 to 347]
  IL-13 -Tetanus toxoid, Day 50: number analyzed (Participants) | 10 | 16
  IL-13 -Tetanus toxoid, Day 50 | 247 [-21.88 to 516] | 293 [94 to 491]

2. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Receiving Two Doses of aTIV and TIV
Description: The number of subjects reporting unsolicited AEs between Day 1 and the study termination i.e., Day 50, after receiving two doses of aTIV and TIV. Data are reported based on the Safety Set.
Time Frame: Day 1 to Day 50 post vaccination
Population: All subjects in the Exposed Set (all enrolled subjects who actually received a study vaccine) who provided post-baseline safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | aTIV Group | TIV Group
Number analyzed (Participants) | 43 | 41
Participants
  Any Adverse Event (AE) | 20 | 18
  At least possibly related AE | 1 | 3
  Any SAE | 0 | 2
  At least possibly related SAE | 0 | 0
  AE leading to discontinuation | 0 | 0
  Death | 0 | 0

3. Secondary Outcome: Percentage of Subjects Achieving Seroconversion or Significant Increase in HI Titer
Description: To evaluate the immune responses by seroconversion of aTIV or TIV according to CHMP criteria for seasonal influenza vaccines as determined by hemagglutination inhibition (HI) test on plasma from previously unvaccinated healthy children aged 6 to < 36 months for all three strains.
  Criteron: The proportion of subjects achieving seroconversion or significant increase in HI titer should be > 40%.
Time Frame: Day 50
Population: Per Protocol Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | aTIV Group | TIV Group
Number analyzed (Participants) | 25 | 30
Percentage of participants
  A/H1N1/California | 100 [86 to 100] | 73 [54 to 88]
  A/H3N2/Victoria | 100 [86 to 100] | 93 [78 to 99]
  B/Brisbane | 100 [86 to 100] | 53 [34 to 72]

4. Secondary Outcome: Geometric Mean Ratios (GMR)
Description: To evaluate the immune responses by mean geometric increase (GMR) of aTIV or TIV according to CHMP criteria for seasonal influenza vaccines as determined by hemagglutination inhibition (HI) test on plasma from previously unvaccinated healthy children aged 6 to < 36 months for all three strains.
  Criterion: Mean geometric increase (GMR) should be > 2.5.
Time Frame: Day 50/Day 1
Population: Per Protocol Set
Measure: Geometric Mean (95% Confidence Interval); unit: titer ratio
Arm/Group | aTIV Group | TIV Group
Number analyzed (Participants) | 25 | 30
titer ratio
  A/H1N1/California | 41 [23 to 74] | 9.99 [5.87 to 17]
  A/H3N2/Victoria | 199 [130 to 303] | 35 [24 to 51]
  B/Brisbane | 34 [22 to 52] | 5.63 [3.83 to 8.29]

5. Secondary Outcome: Percentage of Subjects With HI Titers >1:40
Description: To evaluate the immune responses by proportion of subjects with HI titers >1:40 of aTIV or TIV according to CHMP criteria for seasonal influenza vaccines as determined by hemagglutination inhibition (HI) test on plasma from previously unvaccinated healthy children aged 6 to < 36 months for all three strains.
  Criterion: The proportion of subjects with HI titers >1:40 should be > 70%
Time Frame: Day 50
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | aTIV Group | TIV Group
Number analyzed (Participants) | 25 | 30
Percentage of participants
  A/H1N1/California | 100 [86 to 100] | 93 [78 to 99]
  A/H3N2/Victoria | 100 [86 to 100] | 97 [83 to 100]
  B/Brisbane | 100 [86 to 100] | 57 [37 to 75]

ADVERSE EVENTS:
Time Frame: All solicited AEs and unsolicited AEs were collected from Day 1 to Day 7; all unsolicited SAEs, medically attended AEs, AEs leading to withdrawal from the study were collected from Day 1 to Day 50.
Arm/Group | aTIV (6 to <36 Months) | TIV (6 to <36 Months)
Serious Adverse Events (participants affected / at risk) | 0/43 | 2/41
Other Adverse Events (participants affected / at risk) | 37/43 | 29/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | aTIV (6 to <36 Months) (N=43) | TIV (6 to <36 Months) (N=41)
Varicella (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | aTIV (6 to <36 Months) (N=43) | TIV (6 to <36 Months) (N=41)
Somnolence (Nervous system disorders) | 11 | 12
Crying (General disorders) | 6 | 7
Injection site erythema (General disorders) | 8 | 2
Injection site haemorrhage (General disorders) | 4 | 1
Injection site induration (General disorders) | 3 | 3
Injection site pain (General disorders) | 11 | 9
Pyrexia (General disorders) | 19 | 15
Nasopharyngitis (General disorders) | 5 | 4
Bronchitis (General disorders) | 3 | 1
Eating Disorder (Psychiatric disorders) | 11 | 11
Irratability (Psychiatric disorders) | 11 | 7
Diarrhoea (Gastrointestinal disorders) | 11 | 11
Vomiting (Gastrointestinal disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days